CLINICAL TRIAL: NCT03706820
Title: Hemodynamic Study of the Pulmonary Circulation in Exercise in Patients With Pulmonary Fibrosis
Brief Title: Exercise Hemodynamics in Patients With Pulmonary Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, EVAGGELIA PANAGIOTIDOU, Phd candidate, Resident of Pulmonary medicine, G.H.G.Papanikolaou, Thessaloniki, Greece, Aristotle University Of Thessaloniki
Other Study IDs: MED-AUTH-3.1/02-05-2018
Record Dates: First submitted 2018-09-29; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Exercise Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal rest and exercise hemodynamics
- normal rest and abnormal exercise hemodynamics
- resting pulmonary hypertension
- abnormal wedge pressure at exercise

SUMMARY:
The study evaluates the rest and exercise hemodynamics of patients presenting either idiopathic fibrotic pulmonary disease or pulmonary fibrosis secondary to connective tissue disease.

DETAILED DESCRIPTION:
Patients with fibrotic pulmonary disease of the above origin will undergo detailed assessment of functional status with the following examinations: pulmonary function tests, echocardiogram, 6 minute exercise test, cardiopulmonary exercise test (in the absence of contra-indications) and finally right heart catheterization. Hemodynamic assessment will take place at rest and at exercise following the exercise protocol that was recommended by Herve et al (ERJ 2015) using a cycle ergometer at bedside.

The purposes of the study are:

1. to evaluate the response of the hemodynamic parameters at exercise compared to the resting parameters in this patient group.
2. to discriminate between precapillary from postcapillary etiology of pulmonary hypertension.
3. to correlate non-invasive parameters of functional limitation with invasive hemodynamic parameters.
4. to assess the prognostic role of exercise induced pulmonary hypertension in the specific patient group.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of pulmonary fibrosis secondary to connective tissue disease, according to the American College of Rheumatology/European League Against Rheumatism (ACR-EULAR) revised classification criteria , or diagnosis of idiopathic fibrotic diffuse pulmonary disease according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines
2. Forced vital capacity (FVC) ≥ 40 %

Exclusion Criteria:

1. Presence of contra-indications to exercise tests, such as acute myocardial infarction, unstable angina, uncontrollable arrythmia or skeletal disease that limits the ability to exercise.
2. History of pulmonary embolism during the year before enrollment
3. Presence of severe valvular disease.
4. Current treatment with vasoactive drugs of the pulmonary circulation
5. Pulmonary wedge pressure (PAWP) at rest > 15 mmHg

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are currently followed up in the Respiratory Clinics of the investigator's hospital and will be enrolled if suitable after having signed the form of consent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in total pulmonary resistance (TPR) from rest to exercise | 2nd minute,4th minute, 6th minute, 8th minute
  The patient undergoes right heart catheterization and all hemodynamic variables are measured at rest and at exercise. TPR is derived by the following equation : mean pulmonary artery pressure/ cardiac output (mPAP/CO). TPR is measured at rest and at exercise following a specific protocol. The measurements are made at rest, then at the sequential exercise steps of increasing work resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia G Pitsiou, MD, PhD, Study Chair — Aristotle University Of Thessaloniki
Locations (1):
- G.H. G. Papanikolaou, Thessaloniki, Asvestochori, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kovacs G, Herve P, Barbera JA, Chaouat A, Chemla D, Condliffe R, Garcia G, Grunig E, Howard L, Humbert M, Lau E, Laveneziana P, Lewis GD, Naeije R, Peacock A, Rosenkranz S, Saggar R, Ulrich S, Vizza D, Vonk Noordegraaf A, Olschewski H. An official European Respiratory Society statement: pulmonary haemodynamics during exercise. Eur Respir J. 2017 Nov 22;50(5):1700578. doi: 10.1183/13993003.00578-2017. Print 2017 Nov. PMID 29167297
- [Result] Herve P, Lau EM, Sitbon O, Savale L, Montani D, Godinas L, Lador F, Jais X, Parent F, Gunther S, Humbert M, Simonneau G, Chemla D. Criteria for diagnosis of exercise pulmonary hypertension. Eur Respir J. 2015 Sep;46(3):728-37. doi: 10.1183/09031936.00021915. Epub 2015 May 28. PMID 26022955
- [Derived] Panagiotidou E, Betaoutou A, Fouka E, Papakosta D, Chatzopoulos E, Sourla E, Markopoulou A, Kioumis I, Stanopoulos I, Pitsiou G. Phenotyping exercise limitation of patients with Interstitial Fibrosing Lung Disease: the importance of exercise hemodynamics. Pulmonology. 2024 Mar-Apr;30(2):104-112. doi: 10.1016/j.pulmoe.2022.03.012. Epub 2022 May 11. PMID 35568651